CLINICAL TRIAL: NCT00018343
Title: Alzheimer's Disease and Aging: Therapeutic Potential of Estrogen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGCG-007-97F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Estrogens

INTERVENTIONS:
Drug: estrogen

SUMMARY:
This study is designed to evaluate the potential beneficial effects of estrogen on cognitive function of women with Alzheimer's Disease.

ELIGIBILITY:
* Post menopausal women with alzheimer's disease
* free of any major medical or neurological disease,
* medically safe to be treated with estrogen.

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-04; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, Ph.D; Laura Baker, Ph.D; Murray Raskind, M.D.
Locations (1):
- VA Puget Sound Health Care System, Lakewood, Washington, United States